CLINICAL TRIAL: NCT01833741
Title: A Study of LUMIGAN® RC in the Clinical Setting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLEAR
Record Dates: First submitted 2013-04-15; First posted 2013-04-17 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Glaucoma, Primary Open Angle; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bimatoprost 0.01% (Experimental): Bimatoprost 0.01% (LUMIGAN® RC) administered as one drop in the study eye(s) each evening for 12 weeks.
  Interventions: Drug: Bimatoprost 0.01%

INTERVENTIONS:
Drug: Bimatoprost 0.01% — Bimatoprost 0.01% (LUMIGAN® RC) administered as one drop in the study eye(s) each evening for 12 weeks.
  Other Names: LUMIGAN® RC

SUMMARY:
This study will evaluate bimatoprost 0.01% (LUMIGAN® RC) in patients with elevated intraocular pressure (IOP) due to primary open angle glaucoma (POAG) or ocular hypertension (OHT) in a clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Elevated IOP due to either primary open-angle glaucoma or ocular hypertension
* Determined by the treating physician to require treatment with LUMIGAN® RC

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1137 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Barrie, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bimatoprost 0.01%
Started | 1137
Completed | 997
Not Completed | 140

BASELINE CHARACTERISTICS:
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 1137
Age Continuous [Mean (Standard Deviation); unit: Years] | 66.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 605
  Male | 532

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Treatment-Naive Patients With Ocular Hyperemia
Description: Hyperemia is engorgement of the blood vessels (redness) of the bulbar conjunctiva of the eye (the clear membrane covering the white surface of the eye). Hyperemia is graded on a 5 point scale where 0=none (normal), 0.5=trace (trace flush reddish pink), 1=Mild (mild flush reddish color), 2=Moderate (bright red color) and 3=severe (deep bright diffuse redness). Naive patients did not use glaucoma medication prior to study entry.
Time Frame: Week 12
Population: All patients who were consented and completed the Baseline visit, and who had data for Week 12
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 460
Percentage of Patients
  0 (none) | 32.2
  +0.5 (trace) | 39.8
  +1 (mild) | 21.3
  +2 (moderate) | 5.9
  +3 (severe) | 0.9

2. Secondary Outcome: Percent Change From Baseline in Intraocular Pressure (IOP) in the Study Eye of Treatment-Naive Patients
Description: IOP is a measurement of the fluid pressure inside the eye. Naive patients did not use glaucoma medication prior to study entry. A negative number change from baseline indicates a reduction in IOP (improvement), and a positive number change from baseline indicates an increase (worsening).
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat: all patients who were consented and completed the Baseline visit
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 522
Percent Change | -30.9 (15.4)

3. Secondary Outcome: Percent Change From Baseline in IOP in the Study Eye of Previously Treated (Switched) Patients
Description: IOP is a measurement of the fluid pressure inside the eye. Previously treated patients used glaucoma medication prior to study entry and were switched from their previous therapy to study treatment. A negative number change from baseline indicates a reduction in IOP (improvement), and a positive number change from baseline indicates an increase (worsening).
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat: all patients who were consented and completed the Baseline visit
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 450
Percent Change | -16.1 (18.8)

4. Secondary Outcome: Percent Change From Baseline in IOP in the Study Eye of Patients Treated With Adjunctive Therapy
Description: IOP is a measurement of the fluid pressure inside the eye. Previously treated patients used glaucoma medication prior to study entry and added study treatment as adjunctive therapy. A negative number change from baseline indicates a reduction in IOP (improvement), and a positive number change from baseline indicates an increase (worsening).
Time Frame: Baseline, 12 Weeks
Population: Intent to Treat: all patients who were consented and completed the Baseline visit
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 165
Percent Change | -16.1 (20.4)

5. Secondary Outcome: Change From Baseline in IOP in the Study Eye of Treatment-Naive Patients
Description: IOP is a measurement of the fluid pressure inside the eye. A negative number change from baseline indicates a reduction in IOP (improvement), and a positive number change from baseline indicates an increase (worsening).
Time Frame: Baseline, Week 6, Week 12
Population: Intent to Treat: all patients who were consented and completed the Baseline visit
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 522
Millimeters of Mercury (mmHg)
  Baseline | 23.5 (5.8)
  Change from Baseline at Week 6 | -7.4 (4.9)
  Change from Baseline at Week 12 | -7.7 (4.9)

6. Secondary Outcome: Change From Baseline in IOP in the Study Eye of Previously Treated (Switched) Patients
Description: as for outcome 5
Time Frame: Baseline, Week 6, Week 12
Population: Intent to Treat: all patients who were consented and completed the Baseline visit
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 450
Millimeters of Mercury (mmHg)
  Baseline | 20.3 (4.6)
  Change from Baseline at Week 6 | -3.5 (4.3)
  Change from Baseline at Week 12 | -3.7 (4.3)

7. Secondary Outcome: Change From Baseline in IOP in the Study Eye of Patients Treated With Adjunctive Therapy
Description: as for outcome 5
Time Frame: Baseline, Week 6, Week 12
Population: Intent to Treat: all patients who were consented and completed the Baseline visit
Measure: Mean (Standard Deviation); unit: Millimeters of Mercury (mmHg)
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 165
Millimeters of Mercury (mmHg)
  Baseline | 20.8 (5.2)
  Change from Baseline at Week 6 | -3.8 (4.7)
  Change from Baseline at Week 12 | -3.7 (4.6)

8. Secondary Outcome: Percentage of Patients Discontinuing Due to Ocular Adverse Events
Description: Ocular adverse events are defined as any untoward medical occurrence in a patient's eye(s) during study participation, regardless of relationship to treatment.
Time Frame: 12 Weeks
Population: Intent to Treat: all patients who were consented and completed the Baseline visit
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 1137
Percentage of Patients | 3.9

9. Primary Outcome: Percentage of Previously Treated (Switched) Patients With Ocular Hyperemia
Description: Hyperemia is engorgement of the blood vessels (redness) of the bulbar conjunctiva of the eye (the clear membrane covering the white surface of the eye). Hyperemia is graded on a 5 point scale where 0=none (normal), 0.5=trace (trace flush reddish pink), 1=Mild (mild flush reddish color), 2=Moderate (bright red color) and 3=severe (deep bright diffuse redness). Previously treated patients used glaucoma medication prior to study entry and were switched from their previous therapy to study treatment.
Time Frame: Week 12
Population: All patients who were consented and completed the Baseline visit, and who had data for Week 12
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 400
Percentage of Patients
  0 (none) | 35.5
  +0.5 (trace) | 41.0
  +1 (mild) | 17.3
  +2 (moderate) | 6.0
  +3 (severe) | 0.3

10. Primary Outcome: Percentage of Patients Treated With Adjunctive Therapy With Ocular Hyperemia
Description: Hyperemia is engorgement of the blood vessels (redness) of the bulbar conjunctiva of the eye (the clear membrane covering the white surface of the eye). Hyperemia is graded on a 5 point scale where 0=none (normal), 0.5=trace (trace flush reddish pink), 1=Mild (mild flush reddish color), 2=Moderate (bright red color) and 3=severe (deep bright diffuse redness). Previously treated patients used glaucoma medication prior to study entry and added study treatment as adjunctive therapy.
Time Frame: Week 12
Population: All patients who were consented and completed the Baseline visit, and who had data for Week 12
Measure: Number; unit: Percentage of Patients
Arm/Group | Bimatoprost 0.01%
Number analyzed (Participants) | 141
Percentage of Patients
  0 (none) | 28.4
  +0.5 (trace) | 36.9
  +1 (mild) | 24.1
  +2 (moderate) | 9.2
  +3 (severe) | 1.4

ADVERSE EVENTS:
Arm/Group | Bimatoprost 0.01%
Serious Adverse Events (participants affected / at risk) | 3/1137
Other Adverse Events (participants affected / at risk) | 0/1137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bimatoprost 0.01% (N=1137)
Cerebrovascular Accident (Cardiac disorders) | 1
Malaise (General disorders) | 1
Myocardial Infarction (Cardiac disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.